CLINICAL TRIAL: NCT05766787
Title: The Clinical Performance of Two Reusable Silicone Hydrogel Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CLL949-C024
Record Dates: First submitted 2023-03-01; First posted 2023-03-13 (Actual); Results first posted 2024-06-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-05

CONDITIONS: Refractive Ametropia
Keywords: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- LID022821, then AOHP (Other): Serafilcon A contact lenses worn first, with senofilcon A contact lenses worn second, as randomized. Each study lens type will be worn bilaterally (in both eyes) for approximately 14 days. CLEAR CARE will be used for daily cleaning and disinfection.
  Interventions: Device: Serafilcon A contact lenses; Device: Senofilcon A contact lenses; Device: CLEAR CARE
- AOHP, then LID022821 (Other): Senofilcon A contact lenses worn first, with serafilcon A contact lenses worn second, as randomized. Each study lens type will be worn bilaterally (in both eyes) for approximately 14 days. CLEAR CARE will be used for daily cleaning and disinfection.
  Interventions: Device: Serafilcon A contact lenses; Device: Senofilcon A contact lenses; Device: CLEAR CARE

INTERVENTIONS:
Device: Serafilcon A contact lenses — Reusable silicone hydrogel contact lenses worn during the day and removed at night for cleaning and disinfection
  Other Names: LID022821
Device: Senofilcon A contact lenses — Reusable silicone hydrogel contact lenses worn during the day and removed at night for cleaning and disinfection
  Other Names: ACUVUE OASYS® with HYDRACLEAR® PLUS Technology; AOHP
Device: CLEAR CARE — Hydrogen peroxide based contact lens cleaning and disinfecting solution
  Other Names: CLEAR CARE® Cleaning and Disinfecting Solution

SUMMARY:
The purpose of this study is to assess the clinical performance of two reusable silicone hydrogel contact lenses when worn on a daily wear basis.

DETAILED DESCRIPTION:
In this crossover study, subjects will wear each lens product for approximately 14 days and attend 7 scheduled visits. The expected overall duration of exposure to the study products is approximately 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Successful wear of spherical soft contact lenses in both eyes for a minimum of 5 days per week and 8 hours per day during the past 3 months.
* Best Corrected Visual Acuity (BCVA) of 20/25 Snellen (0.10 logMAR) or better in each eye.
* Willing to stop wearing habitual contact lenses for the duration of study participation.
* Other protocol-specific inclusion criteria may apply.

Exclusion Criteria:

* Any eye infection, inflammation, abnormality or disease (including systemic) that contraindicates contact lens wear, as determined by the investigator.
* Any use of systemic or ocular medications for which contact lens wear could be contraindicated, as determined by the investigator.
* Habitual wear of AOHP contact lenses.
* Habitual wear of any daily disposable contact lenses.
* Other protocol-specified exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2023-03-29 (Actual); Primary Completion 2023-06-02 (Actual); Study Completion 2023-06-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Lead Alcon Vision Care, Study Director — Alcon Research, LLC
Locations (15):
- United States (15):
  - Kurata Eyecare Center, Los Angeles, California
  - Dr. Elsa Pao, OD, Oakland, California
  - Pacific Rims Optometry, San Francisco, California
  - Omega Vision Center P.A., Longwood, Florida
  - Kindred Optics at Maitland Vision, Maitland, Florida
  - Vision Health Institute, Orlando, Florida
  - Tallahassee Eye Center, Tallahassee, Florida
  - Heart of America Eye Care, Shawnee Mission, Kansas
  - The Eye Doctors Inc, Eden Prairie, Minnesota
  - Complete Eye Care of Medina, Medina, Minnesota
  - SUNY College of Optometry Clinical Vision Research Center, New York, New York
  - ProCare Vision Centers, Inc., Granville, Ohio
  - West Bay Eye Associates, Warwick, Rhode Island
  - Optometry Group, PLLC, Memphis, Tennessee
  - Total Eye Care PA, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 15 investigative sites located in the United States.
Pre-assignment Details: Of the 190 enrolled, 3 participants were exited prior to randomization as screen failures. Of the 187 randomized, 1 participant was discontinued prior to exposure to the study lenses due to ocular pre-treatment adverse events. This reporting group includes all participants exposed to any study lenses (186).
Units Other Than Participants: eyes
Groups:
- LID022821, Then AOHP: Serafilcon A contact lenses worn first, with senofilcon A contact lenses worn second, as randomized. Each study lens type was worn bilaterally (in both eyes) for approximately 14 days. CLEAR CARE was used for daily cleaning and disinfection.
- AOHP, Then LID022821: Senofilcon A contact lenses worn first, with serafilcon A contact lenses worn second, as randomized. Each study lens type was worn bilaterally (in both eyes) for approximately 14 days. CLEAR CARE was used for daily cleaning and disinfection.
Period: First Wear Period, Approximately 7 Days
Arm/Group | LID022821, Then AOHP | AOHP, Then LID022821
Started | 94; 188 eyes | 92; 184 eyes
Completed | 93; 186 eyes | 89; 178 eyes
Not Completed | 1; 2 eyes | 3; 6 eyes
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 1 | 2
Period: Second Wear Period, Approximately 7 Days
Arm/Group | LID022821, Then AOHP | AOHP, Then LID022821
Started | 93; 186 eyes | 88; 176 eyes (One subject was discontinued between first and second period due to Physician decision.)
Completed | 93; 186 eyes | 87; 174 eyes
Not Completed | 0; 0 eyes | 1; 2 eyes
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set: All randomized subjects who are exposed to any study lenses evaluated in this study.
Groups:
- Total: Total of all reporting groups
Arm/Group | LID022821, Then AOHP | AOHP, Then LID022821 | Total
Number analyzed (Participants) | 94 | 92 | 186
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.1 (8.6) | 33.9 (9.0) | 34.0 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 64 | 124
  Male | 34 | 28 | 62
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 66 | 62 | 128
  Black or African American | 7 | 9 | 16
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 20 | 19 | 39
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Other | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 7 | 13
  Not Hispanic or Latino | 88 | 85 | 173

OUTCOME MEASURES:

1. Primary Outcome: Least Squares Mean Distance VA With Study Lenses at Week 1
Description: Visual acuity (VA) was assessed for each eye individually with study lenses in place using logarithmic of the Minimum Angle of Resolution (logMAR) reading charts. LogMAR values typically range from -0.3 (20/10 vision on the Snellen chart) to 1 (20/200 vision). A logMAR acuity of 0.0 corresponds to 20/20 Snellen acuity (normal distance visual acuity), with a negative value denoting better than 20/20 visual acuity.
Time Frame: Week 1 of each lens product worn during the corresponding crossover period
Population: Full Analysis Set: All randomized subjects who were exposed to any study lenses evaluated in this study with data at Week 1 visit.
Measure: Least Squares Mean (Standard Error); unit: logMAR
Units Other Than Participants: eyes
Groups:
- LID022821: Serafilcon A contact lenses worn first or second, as randomized, in both eyes for approximately 14 days. CLEAR CARE was used for daily cleaning and disinfection.
- AOHP: Senofilcon A contact lenses worn first or second, as randomized, in both eyes for approximately 14 days. CLEAR CARE was used for daily cleaning and disinfection.
Arm/Group | LID022821 | AOHP
Number analyzed (Participants) | 181 | 185
Number analyzed (eyes) | 362 | 370
logMAR | -0.11 (0.005) | -0.10 (0.005)
Statistical Analysis 1: Comparison: LID022821 vs AOHP; Test type: Non-Inferiority — Noninferiority in distance VA was declared if upper confidence limit was less than 0.05; Since a noninferiority hypothesis is being tested, a p-value is not applicable. Confidence limit is being reported and compared to the noninferiority margin; Least Squares Mean Difference = -0.01, 95% CI 1-sided [upper limit -0.01], Standard Error of Mean 0.003 — LSM results based on mixed effects repeated measures model with both fixed (lens, period, sequence, visit, and lens by visit interaction) and random (subject) effects. Difference = LID022821 minus AOHG. Sign is retained with the rounded value

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from time of consent to study exit, approximately 28 days.
Description: AEs were obtained through solicited and spontaneous comments from subjects and through observations by the Investigator. "At Risk" population for ocular AEs is reported in units of eyes; all other populations are reported in units of subjects. This analysis population includes all subjects/eyes exposed to any study lenses, as treated. The Other (Not Including Serious) Adverse Event table reports only the AEs that occurred above a 5% threshold in one or more arms.
Groups:
- Pretreatment: Events reported in this group occurred prior to exposure to the study contact lenses.
- LID022821 - Ocular; LID022821 - Non-Ocular: Events reported in this group occurred while exposed to the serafilcon A contact lenses.
- AOHP - Ocular; AOHP - Non-Ocular: Events reported in this group occurred while exposed to the senofilcon A contact lenses.
Arm/Group | Pretreatment | LID022821 - Ocular | LID022821 - Non-Ocular | AOHP - Ocular | AOHP - Non-Ocular
All-Cause Mortality (participants affected / at risk) | 0/186 | 0/364 | 0/182 | 0/370 | 0/185
Serious Adverse Events (participants affected / at risk) | 0/186 | 0/364 | 0/182 | 0/370 | 0/185
Other Adverse Events (participants affected / at risk) | 0/186 | 0/364 | 0/182 | 0/370 | 0/185

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.

DOCUMENTS (2):
  • Study Protocol (2023-04-13): https://cdn.clinicaltrials.gov/large-docs/87/NCT05766787/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-03): https://cdn.clinicaltrials.gov/large-docs/87/NCT05766787/SAP_001.pdf